CLINICAL TRIAL: NCT01234870
Title: Comprehensive Evaluation of Ischemic Heart Disease Using MRI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, James Carr, Director of Cardiovascular Imaging, Department of Radiology,Associate Professor of Radiology and Medicine, Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR1_STU00006013; ASCA-9J02 (Other Grant/Funding Number: Astellas Pharma Global Development, Inc)
Record Dates: First submitted 2010-10-05; First posted 2010-11-04 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Heart Disease, Ischemic; Atherosclerosis, Coronary
Keywords: Myocardial Perfusion Imaging; Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease | interventions — Gadolinium; Gadolinium DTPA; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ischemic heart disease patients (Experimental): Patients with suspected ischemic heart disease prospectively recruited for first pass myocardial perfusion MRI. All subject to receive Gadolinium infusion of 0.075 mmol/kg at rate of 4 ml/sec. Adenosine administered at a rate of 0.14 mg/kg/min for a duration of 4 minutes to induce stress.
  Interventions: Drug: Gadolinium; Drug: Adenosine

INTERVENTIONS:
Drug: Gadolinium
  Other Names: Magnevist, Bayer HealthCare Pharmaceuticals
Drug: Adenosine

SUMMARY:
The purpose of the study is to assess the diagnostic performance of fully automated motion corrected (MC) first pass myocardial perfusion MRI, compared to the original non-corrected first pass myocardial perfusion images in a cohort of patients with suspected ischemic heart disease, using coronary angiography as the reference standard. It is expected that this improved comprehensive protocol for cardiac MRI be accurate at detecting significant coronary artery disease and may obviate the need for other more expensive and invasive diagnostic tests currently used.

DETAILED DESCRIPTION:
Coronary heart disease is the leading cause of death and disability in the US, accounting for about one-third of all deaths in subjects over age 35.

With the development of newer Magnetic Resonance Imaging (MRI) techniques, such as faster pulse sequences and parallel imaging, cardiac MRI has become a routine tool for the evaluation and detection of myocardial ischemic disease. First pass myocardial perfusion (FPMP) using MRI is increasingly being used to assess ischemic heart disease. MRI offers the advantages of spatial resolution sufficient to differentiate between subendocardial and subepicardial perfusion; shorter examination time and also lack of ionizing radiation. Left ventricle cine gradient echo imaging can be used to assess regional ventricular function. Left ventricular myocardial viability can also be easily assessed at the same time in order to determine the amount of viable left ventricular myocardium and the percentage of irreversibly scarred myocardium by delayed enhanced images. Viability imaging is usually added to the perfusion protocol to increase specificity by allowing detection of fixed perfusion defects, which represent scar. The ultimate cardiac MRI protocol would be to combine both of these imaging strategies with a reliable and accurate coronary Magnetic Resonance Angiography(MRA) technique, such that obstructive coronary artery disease could be evaluated comprehensively at the same time. If all of these techniques can be combined together in a single study, it may be feasible to finally achieve a "one stop shop" for cardiac Magnetic Resonance Imaging.

ELIGIBILITY:
Inclusion Criteria:

Under an Institutional Committee on Human Research board approved protocol 80 patients with a suspected myocardial ischemic disease recruited from the cardiac cath laboratory will be recruited in this prospective study. Volunteers will be recruited for the purpose of protocol development and will not be included in analysis. All subjects will be screened for glomerular filtration rate (GFR) within 24 hours before the exam. All patients must have a GFR > 30 mL/min/1.73m2 to be part of the study.

All subjects will be selected following the Nephrogenic Systemic Fibrosis (NSF) guidelines. All dialysis patients or end-stage renal disease patients with a creatinine clearance of < 30 mL/min will not be selected for the study to avoid NSF. Patients with GFR < 60 ml/min but >30 ml/min will receive a reduced dose of Gadolinium contrast (0.1 ml/kg).

Exclusion Criteria:

1. Age <18 years;
2. Known contraindication to MR imaging (such as pacemaker placement, magnetic implants, etc);
3. Claustrophobia;
4. Inability to perform an adequate breath-hold for imaging,
5. Inability to provide informed consent;
6. all subjects will be will be screened for GFR within 24 hours before the exam and subjects presenting with GFR < 30 ml/min will be excluded;
7. Pregnant and lactating women;
8. Patients with hypersensitivity to gadolinium contrast agents, metoprolol, adenosine, or nitroglycerin;
9. Contra indication for Adenosine

   1. 2nd- or 3rd-degree atrioventricular block (except in patients with a functioning artificial pacemaker)
   2. Sinus node disease (except in patients with a functioning artificial

      pacemaker)
   3. Unstable angina
   4. Acute myocardial infarction
   5. Known or suspected bronchoconstrictive or bronchospastic lung

      disease (e.g., asthma)
   6. Hypersensitivity to adenosine
   7. Caffeine within 12-24 hours
   8. Theophylline and Dipyridamole products within 24 hours.
10. Contra indication for Metoprolol

    1. sinus bradycardia
    2. heart block greater than first degree
    3. Cardiac Failure
    4. Bronchospastic Disease
11. Contra indication for Nitroglycerin

    1. Early myocardial infarction, severe anemia, increased intracranial pressure, and those with a known hypersensitivity to nitroglycerin.

b .Administration of Nitrostat (nitroglycerin tablets, USP) is contraindicated in patients who are using Viagra® since Viagra has been shown to potentiate the hypotensive effects of organic nitrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Carr, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ischemic Heart Disease Patients
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 40 patients were successfully scanned per the imaging protocol and all images collected were of diagnostic quality and successfully processed. Age, gender, race, ethnicity and BMI were collected on all 40 patients and all have been included in the analyses.
Groups:
- Adenosine: Adenosine (Adenoscan) will be infused intravenously at a dose of 0.14mg/kg/min for a total of 4 mins.
  adenosine: Adenosine will be infused intravenously at a dose of 0.14mg/kg/min for a total of 4 mins
Arm/Group | Adenosine
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 30
  More than one race | 0
  Unknown or Not Reported | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.57 (5.83)

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Image Quality Rating
Description: The purpose of the study is to assess the incremental value of diagnostic performance using a fully-automated, motion-corrected (MC) first pass myocardial perfusion image acquisition protocol compared to images obtained under a non-corrected, breath-hold, shallow-breathing first pass myocardial perfusion image acquisition protocol in patients with suspected ischemic heart disease. The MR images resulting from two different image acquisition techniques, including Non-Corrected Breath-Hold Shallow-Breathing and Motion-Corrected, were assessed independently by two radiologists (average of 7 years of experience in reading cardiac MRI) using the American Heart Association modified 16 segment model and were evaluated using a four point Likert scale (1 = poor, 2 = fair, 3 = good, and 4 = excellent) for image quality
Time Frame: Cross sectional study; magnetic resonance images were obtained on all patients using two different acquisition methods.
Measure: Mean (Standard Deviation); unit: units on a likert scale
Arm/Group | Ischemic Heart Disease Patients
Number analyzed (Participants) | 40
units on a likert scale
  Motion Corrected Images | 3.57 (0.66)
  Non-Corrected Breath-Hold, Shallow-Breathing Image | 2.55 (0.81)
Statistical Analysis 1: Comparison: Ischemic Heart Disease Patients; The MR images resulting from two different image acquisition techniques, including Non-Corrected Breath-Hold Shallow-Breathing and Motion-Corrected, were assessed independently by two radiologists (average of 7 years of experience in reading cardiac MRI) using the American Heart Association modified 16 segment model and were evaluated using a four point Likert scale (1 = poor, 2 = fair, 3 = good, and 4 = excellent) for image quality; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Adverse Events to Demonstrate Feasibility of a Comprehensive Cardiac Magnetic Resonance Imaging Protocol
Description: Adverse events relating to administration of adenosine during a coronary heart disease comprehensive cardiac MRI study.
Time Frame: 14 days
Measure: Number; unit: occurances of adverse events
Arm/Group | Adenosine
Number analyzed (Participants) | 40
occurances of adverse events | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for 14 days following administration of adenosine.
Description: Patients were monitored for adverse events on the day of the MR scan. Following administration of adenosine for stress testing, patients were monitored until fifteen minutes after patient vitals returned to baseline. Following the day of participation, patients were monitored for any serious adverse experiences for 14 days.
Arm/Group | Adenosine
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
The small number of subjects results in reduced statistical power; The cohort was selected from patients at a single medical center, potentially reducing generalizability; Variability in patient behavior during MR scans may affect analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No